CLINICAL TRIAL: NCT00989326
Title: Comparative Follow-up Schedule With Home Monitoring
Brief Title: Evaluate the Benefits of Pacemaker Follow-Up With Home-Monitoring
Acronym: COMPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik France (Industry)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Nicolas Canot, Biotronik France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HS037
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2009-10

CONDITIONS: Pacemaker, Artificial; Bradycardia
Keywords: Remote monitoring; Pacemaker; Follow up; Follow-up studies
MeSH Terms: conditions — Bradycardia | interventions — Blood Glucose Self-Monitoring; Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CONTROL group (Active Comparator): The patients receive standard of care for 18 months. The CONTROL group patients will be equipped with Home Monitoring. However, the Home Monitoring data will not be used for patient surveillance; i. e. the patient will be followed in the conventional manner.
  Interventions: Other: Home Monitoring
- ACTIVE group (Experimental): The patients are followed by Home monitoring only. Every patient must be seen by his physician 18 months after enrolment for regular follow-up. Within this period, the additional Pace Maker follow-up or therapeutic intervention will be primarily triggered on cardio-reports reception or patient/physician call
  Interventions: Other: Home Monitoring

INTERVENTIONS:
Other: Home Monitoring — Both patient groups are followed for 18 months and will be followed with Home Monitoring switched on. The data from the CONTROL group will not be presented online to the attending physician, but a retrospective analysis on differences between the two groups will be performed.
  Other Names: Remote monitoring

SUMMARY:
The study investigates whether home monitoring follow-up of Pace-Maker patients is as efficient as conventional method in terms of Significant Serious Adverse Event (SSAE).

DETAILED DESCRIPTION:
Due to its integrated long-distance telemetry, the implantable pacemaker Philos II DR-T is capable of periodically transmitting data from the pacemaker memory to the BIOTRONIK Service Center via patient device. The BIOTRONIK Service Center decodes the data and presents it to the physician on a password secured internet site. Additionally, in case certain event criteria are met, the most important Home Monitoring information are immediately faxed to the physician as an Event Report. These events can be customised by the physician. Thus, the physician will be able to closely monitor the patient and check the adequacy and efficiency of the pacemaker therapy without requiring the patient to visit the physician. The transmitted data comprise information on atrial and ventricular rhythm, atrioventricular conduction and system status.

The purpose of the national prospective, randomized, multicentric clinical study "COMPArative follow-up Schedule with home monitoring" (COMPAS) described here is to evaluate the benefits of pacemaker follow-up with home monitoring in France. The standard follow-up or therapeutic intervention will be deemed based on faxed event Reports reception and Cardio reports analysis on internet site. During the clinical study, the incidence of serious adverse events (hospitalisation, pacemaker dysfunction, and cardiovascular events), economic impact, safety, and practicability will be analysed. The findings from the ACTIVE group will be compared to those of a group receiving standard of care (CONTROL group). Both patient groups are followed for 18 months and will be followed with Home Monitoring switched on. The data from the CONTROL group will not be presented online to the attending physician, but a retrospective analysis on differences between the two groups will be performed.

The trial will be conducted as a prospective, randomised, open, multicenter, national clinical trial. The enrollment of 400 patients in 50 clinical centres in France is anticipated. The principal inclusion criterion is indication for dual chamber pacemaker/ICD implantation. Main exclusion criteria comprise pacemaker dependency.

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing and able to comply with the protocol
* The patient has provided written informed consent
* Patient whose medical situation is stable
* Patient with PHILOS II DR-T Pacemaker >= one month with A/V bipolar lead
* No change of residence expected during study

Exclusion Criteria:

* Spontaneous Ventricular Rhythm < 30 ppm
* Heart failure no controlled by medical treatment
* Post cardiac surgery (< 1 month)
* Post myocardial infarction (< 1 month)
* More than two cardioversion shocks for last 6 month
* A/V Lead dislodgement, or/and impedance, threshold, or sensing failure
* Pocket hematoma with needed intervention
* Pneumothorax / Hemothorax
* Infection
* Automatic Ventricular Threshold Test cannot be realised
* Patient unable to handle Home Monitoring system correctly
* Insufficient GSM coverage at patient's home
* Participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2005-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with serious adverse events detected during and at the end of an 18 months follow-up period is compared for the two groups | 18 months

SECONDARY OUTCOMES:
Efficacy of Home Monitoring to detect pacemaker dysfunction | 18 months
Reduction of associated cost | 18 months
Delay of Home Monitoring to manage adverse events | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe P MABO, Pr, Dr, Principal Investigator — CHU Pontchaillou de Rennes
Locations (1):
- CHU Pontchaillou de Rennes, Rennes, France

REFERENCES:
- [Derived] Mabo P, Victor F, Bazin P, Ahres S, Babuty D, Da Costa A, Binet D, Daubert JC; COMPAS Trial Investigators. A randomized trial of long-term remote monitoring of pacemaker recipients (the COMPAS trial). Eur Heart J. 2012 May;33(9):1105-11. doi: 10.1093/eurheartj/ehr419. Epub 2011 Nov 29. PMID 22127418